CLINICAL TRIAL: NCT01115075
Title: Oscillations in Dietary Fat Intake and Leptin Changes Among People Who Record Dietary Intake Accurately: the Dietitian Study II
Brief Title: Oscillations of Dietary Fat/Carbohydrate Intake Over Interval of 3 to 4 Days
Acronym: Dietitian II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pennington Biomedical Research Center (Other)
Responsible Party: Principal Investigator, George A. Bray, Principal Investigator, Pennington Biomedical Research Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBRC 29017
Record Dates: First submitted 2010-04-14; First posted 2010-05-04 (Estimated); Last update posted 2016-01-25 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
Keywords: Leptin; Changes in leptin may precede the; phasing of oscillations of dietary fat intake
MeSH Terms: interventions — Nutritionists

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dietitian (Experimental): Recruitment of dietitians and senior level or graduate level dietetics students who are not restrained eaters. This group is skilled in identifying and accurately recording food than individuals not trained in dietetics.
  Interventions: Other: Dietary fat/intake of carbohydrate; Behavioral: Spontaneous oscillations of dietary fat/intake of carbohydrate in relation to energy intake.

INTERVENTIONS:
Other: Dietary fat/intake of carbohydrate — Spontaneous intake of fat, carbohydrate, protein and alcohol each day for 17 days.
  Other Names: Dietitian II
Behavioral: Spontaneous oscillations of dietary fat/intake of carbohydrate in relation to energy intake. — Dietitians and senior level or graduate level dietetics students who are not restrained eaters to participate in food intake over 17 days. During this same time interval, integrated energy expenditure will be recorded using doubly-labeled water and day to day energy expenditure by accelerometer. Periodic blood sampling for leptin will be done completed at site intervals.

SUMMARY:
The purpose of this study is to understand the mechanisms for oscillations of dietary fat/carbohydrate intake and how fat intake affect insulin resistance and liver fat over interval of 3 to 4 days.

DETAILED DESCRIPTION:
You will be expected to keep diet records for 17 consecutive days. You will start with a fasting screening visit (only water allowed). A physical exam and Medical history it taken at screening visit. Your body composition will be gathered by CT and Dexa Scan. Blood and urine will be collected for a chemical profile and other determinations. Questionnaires will be administered along with an accelerometer to be worn for the remainder of the study. The final day you will return the dietary records, accelerometer, and a few procedures will be performed as weight.

ELIGIBILITY:
Inclusion Criteria:

* You are a dietitian or a senior level or graduate level dietetics student
* You are between the ages of 21-55 years inclusive and a nonsmoker
* you are not a restrictive diet or strenuous exercise regimen
* You typically eat several meals per day

Exclusion Criteria:

* You have an eating disorder or history
* You abuse alcohol or other substances, and consume no more than 3 alcoholic drinks per day
* You have no current regular use of some over-the-counter medication or prescription medication, excluding headache medicines, blood pressure medications, etc.
* You have gained/lost more than 10 pounds of body weight in the last year
* You have recently had or anticipating significant life changes during the course of your participation in the study.
* You have an eating disorder or history
* You have a major psychiatric illness or history
* You have no serious current clinical disease or surgical condition that may interfere with the study.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2010-03; Primary Completion 2011-03 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Mechanisms for oscillations of dietary fat/carbohydrate intake | 17 consecutive days (11 visits on site)
  Test the spontaneous intake of fat, carbohydrate,protein and alcohol each day for 17 consecutive days. Examine spontaneous oscillations of dietary fat/intake of carbohydrate in relation to energy intake.

SECONDARY OUTCOMES:
Energy Intake | 17 days
  During the same time interval, integrated energy expenditure will be recoreded using doubly-labeled water and day to day energy expenditure by accelerometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Pennington Biomedical Research Center, Baton Rouge, Louisiana, United States